CLINICAL TRIAL: NCT04559984
Title: A Randomized, Multicenter, "No-Treatment" Control Study to Evaluate the Safety and Effectiveness of JUVÉDERM VOLUX® Injectable Gel for the Enhancement of the Chin to Correct Moderate to Severe Retrusion in Chinese Adults
Brief Title: JUVÉDERM VOLUX® for Chin Retrusion in China
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1868-701-008
Record Dates: First submitted 2020-09-17; First posted 2020-09-23 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Chin Retrusion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- JUVÉDERM VOLUX® (Experimental): Participants will be treated with VOLUX XC hyaluronic acid (HA) injectable gel on day 1 with an optional touch-up treatment at week 4 if agreed upon by both the participant and Treating Investigator.
  Interventions: Device: JUVÉDERM VOLUX®
- Control- No treatment (Other): No-treatment during the control period. Optional delayed-treatment with VOLUX XC (initial with optional touch-up) during the Post-Control period.
  Interventions: Device: JUVÉDERM VOLUX®

INTERVENTIONS:
Device: JUVÉDERM VOLUX® — JUVÉDERM VOLUX® injectable gel

SUMMARY:
The objective of this study is to evaluate the safety and effectiveness of JUVÉDERM VOLUX® to correct moderate to severe chin retrusion in Chinese adults.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be at least 18 years of age at the time of signing the ICF
* Male and female
* Participants of Chinese descent
* Participants seeking improvement of chin retrusion
* Chin retrusion (G-Sn-Pog angle of < 172.5°) based on calculations of facial angle derived from digital images obtained using Canfield imaging equipment and software
* Has moderate to severe chin retrusion on the CACRS as determined by EI 2D image evaluation
* Has a reasonable goal for aesthetic improvement in chin retrusion and is able to achieve a 1-point improvement in CACRS score with study intervention in the judgment of TI
* Capable of giving signed informed consent as described in Appendix 10.1.3, which includes compliance with the requirements and restrictions listed in the ICF and in this protocol
* Written informed consent from the participant has been obtained prior to any study-related procedures
* Written documentation has been obtained in accordance with the relevant country and local privacy requirements, where applicable

Exclusion Criteria:

* History of tendency to develop hypertrophic scarring
* History of anaphylaxis or allergy to lidocaine (or any amide-based anesthetics), HA products, or streptococcal protein
* Active autoimmune disease
* Current cutaneous inflammatory or infectious processes (eg, acne, herpes), abscess, an unhealed wound, or a cancerous or precancerous lesion in the chin area (participants with a history of recurrent oral herpes are eligible if prophylactic antiviral/herpes medication is administered for 2 days before study intervention)
* Impaired cardiac conduction, impaired hepatic function, or impaired renal function according to the judgment of the TI based on medical history, laboratory testing results, and other clinical signs and symptoms
* Prior chin or jaw surgery, including cartilage grafts or implantation of any biomaterials
* Permanent dermal filler injected below the subnasale
* Semi-permanent dermal filler or fat injected below the subnasale within 36 months before enrollment
* Temporary dermal filler injected below the subnasale within 12 months before enrollment
* Orthodontics procedures within 12 months before enrollment
* Botulinum toxin treatment in the chin area within 6 months before enrollment
* Mesotherapy or cosmetic facial procedures (eg, face-lift, brow lift, facial reconstructive surgery, laser, photomodulation, intense pulsed light, radio frequency, dermabrasion, moderate or greater depth chemical peel, or other ablative procedures) below the subnasale within 6 months before enrollment
* Current enrollment in an investigational drug or device study or participation in such a study within 30 days before enrollment
* Abnormal and clinically significant results according to the TI or designee, on hematology, clinical chemistry, or urinalysis
* Females who are pregnant, nursing, or planning a pregnancy during the study
* Tattoos, piercings or scars that would interfere with study visual assessments and 3D measurements of chin area in the judgment of TI
* Trauma to the chin or has residual deficiencies, congenital deformities, or scarring which would impact the trial data evaluation in the judgment of TI
* Menstruation at the time of study intervention (study intervention may be delayed as necessary to accommodate menstrual period cessation)
* The participant has a condition or is in a situation which, in the TI's opinion, may put the participant at significant risk, may confound the study results, or may interfere significantly with the participant's participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2022-08-26 (Actual); Study Completion 2022-08-26 (Actual)

PRIMARY OUTCOMES:
Change from baseline in glabella-subnasale-pogonion (G-Sn-Pog) angle at Week 24 | Change from Baseline to Week 24
  The G-Sn-Pog angle is the angle formed by the point on the glabella, subnasale, and pogonion.

SECONDARY OUTCOMES:
China (Allergan) Chin Retrusion Scale (CACRS) responder status based on the Evaluating Investigator's (EI) assessment of 2D images at Week 24 | Week 24
  The CACRS is a validated 5-point ordinal scale developed by Allergan to grade the severity of chin retrusion. The scale ranges from 0=none to 4=severe.
Overall scores of Satisfaction with Chin module of the FACE-Q questionnaire at Week 24 | Week 24
  The subject will assess satisfaction using the 10 items on the Satisfaction with Chin FACE-Q.
Responder status for participant and EI assessments of global aesthetic improvement in the chin and jaw area using the Global Aesthetic Improvement Scale (GAIS) at Week 24 | Week 24
  The GAIS is a 5-point scale where: 2=much improved, 1=improved, 0=no change, -1=worse and -2=much worse.
Number of patients experiencing one or more treatment emergent adverse events (TEAEs) | Up to week 52
  The number of patients who experienced one or more TEAEs

CONTACTS AND LOCATIONS:
Overall Officials: ALLERGAN INC., Study Director — Allergan
Locations (7):
- China (7):
  - Plastic Surgery Hospital(Institute), Cams, Pumc /ID# 224441, Beijing, Beijing Municipality
  - Beijing Hospital /ID# 224440, Beijing, Beijing Municipality
  - Nanfang Hospital of Southern Medical University /ID# 224442, Guangzhou, Guangdong
  - Union Hospital Tongji Medical College Huazhong University of Science and Technol /ID# 224444, Wuhan, Hubei
  - Nanjing Drum Tower Hospital /ID# 224439, Nanjing, Jiangsu
  - Peking University International Hospital /ID# 224438, Beijing
  - Shanghai Ninth People's Hospital,Shanghai Jiaotong University School of Medicine /ID# 224445, Shanghai

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols, analyses plans, clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous independent scientific research, and will be provided following review and approval of a research proposal and statistical analysis plan and execution of a data sharing statement. Data requests can be submitted at any time after approval in the US and/or EU and a primary manuscript is accepted for publication. For more information on the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: clinical study report synopsis — https://www.abbvieclinicaltrials.com/study/?id=1868-701-008#additional-resources-section